CLINICAL TRIAL: NCT07045454
Title: A Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of MHB118C Injection in Patients With Advanced Solid Tumors
Brief Title: A Study of MHB118C Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHB118C-A-101
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Advanced Malignant Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHB118C for Injection (Experimental): MHB118C for Injection Q3W
  Interventions: Drug: MHB118C for Injection

INTERVENTIONS:
Drug: MHB118C for Injection — IV administration by Q3W; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.

SUMMARY:
This is a first-in-human, open-label, multicenter Phase I study of MHB118C in patients with advanced solid tumors. The study was designed to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of MHB118C monotherapy.

DETAILED DESCRIPTION:
This first-in-human clinical trial of MHB118C comprises two parts: a dose escalation phase and indication expansion phase. The dose escalation phase is an open-label, multicenter study including dose escalation and PK expansion cohorts. The primary objectives are to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of MHB118C in patients with advanced solid tumors, and to determine the maximum tolerated dose (MTD). In this phase, additional patients may be enrolled in the PK expansion part at dose levels that have completed DLT (dose-limiting toxicity) evaluation.

Based on the safety, PK, and preliminary efficacy data from the completed DLT-evaluated dose levels, the sponsor will initiate the indication expansion phase. This phase is an open-label, multicenter, multi-cohort study designed to further evaluate the safety and efficacy of MHB118C monotherapy in patients with specific types of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agrees to participate in the study and signs the informed consent form.
2. Age ≥ 18 years, no restriction on gender.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Estimated life expectancy ≥ 3 months.
5. Able to understand and comply with the study protocol and follow-up procedures.
6. Histologically or cytologically confirmed advanced solid tumors that are refractory to standard therapy, intolerant to standard therapy, or have no standard treatment options.
7. At least one measurable lesion per RECIST v1.1 criteria.
8. Adequate organ function.

Exclusion Criteria:

1. History of ≥2 primary malignancies within 5 years prior to informed consent.
2. Received chemotherapy within 3 weeks, radiotherapy within 4 weeks (2 weeks for palliative bone radiotherapy), or biologic, endocrine, or immunotherapy within 4 weeks before first study dose.
3. Brain metastases, leptomeningeal disease, brainstem metastases, or spinal cord compression.
4. Severe lung disease affecting pulmonary function.
5. Active systemic infection requiring treatment within 7 days before dosing.
6. Serious cardiovascular or cerebrovascular diseases
7. Uncontrolled third-space effusions not suitable for enrollment.
8. Known hypersensitivity or delayed allergic reaction to the investigational product or its components.
9. Drug abuse or other medical/psychiatric condition that may interfere with study participation or results.
10. Known alcohol or drug dependence.
11. Pregnant or breastfeeding women, or individuals planning to conceive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) for MHB118C | Up to day 21 from the first dose
  DLTs will be assessed during the dose-escalation phase and are defined as toxicities related to MHB118C
Maximum tolerated dose (MTD) for MHB118C | Up to day 21 from the first dose
  To determine the MTD for further evaluation of IV administration of MHB118C in subjects with advanced solid tumors.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Baseline up to 5 years
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0].
Pharmacokinetic (PK) parameters of total antibody, ADC, and free toxin at various time points | Baseline up to 5 years
  The PK parameters at different time points include:Area Under the Concentration-Time Curve (AUC)
Immunogenicity | Baseline up to 5 years
  Proportion of subjects who develop anti-MHB118C antibodies (ADA).
ORR determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline. ORR is evaluated by the number of participants with best overall response of CR and PR .
Duration of response (DOR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  DoR was defined as the period from the first occurrence of CR or PR to PD or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used.
Disease control rate (DCR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline. DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD).
Progression-free survival (PFS) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline. PFS was defined as the time from random assignment (dose expansion stage) or first dose (dose escalation stage) to PD or death from any cause.
Overall survival (OS) | Baseline up until death up to approximately 5 years
  OS was defined as the time from random assignment or first dose to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No